CLINICAL TRIAL: NCT05680220
Title: A Double-blinded, Randomized Placebo-controlled Trial of 40 Hz Light Neurostimulation Therapy for Patients With Depression
Brief Title: 40 Hz Light Neurostimulation for Patients With Depression (FELIX)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Martiny (Other)
Collaborators: Technical University of Denmark (Other); OptoCeutics (Industry)
Responsible Party: Sponsor-Investigator, Klaus Martiny, Professor, Head of NID-Group, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Organization: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FELIX
Record Dates: First submitted 2023-01-03; First posted 2023-01-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: 40 Hz stimulation; Major Depressive Disorder; Light therapy; GENUS
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Neurostimulation System (NSS) (Experimental): Exposure to the NSS device set to 40 Hz invisible spectral flicker 1 hour a day
- Sham Neurostimulation System (NSS) (Placebo Comparator): Exposure to the NSS device set to continuous color-matched white light for 1 hour a day

INTERVENTIONS:
Device: Neurostimulation System (NSS): Active Setting — Exposure to the active device for 1 hour a day for 6 weeks
Device: Neurostimulation System (NSS): Sham Setting — Exposure to the sham device for 1 hour a day for 6 weeks

SUMMARY:
Recent research in mice models of Alzheimer's disease (AD) has demonstrated that one hour per day of exposure to 40 Hz flickering light therapy can halt the disease's progression, and improve cognition and memory. Moreover, recent data suggest that 40 Hz light stimulation may induce neuroplasticity and reduce neuroinflammation.

In this study, the investigators aim to evaluate the antidepressant effects of 40 Hz light stimulation in Major Depressive Disorder (MDD). Patients will be exposed to 40 Hz invisible spectral flickering light (active setting) or continuous non-flickering white light (sham setting) in a home setting for 1 hour each day.

DETAILED DESCRIPTION:
Major depression is a major societal challenge worldwide and a substantial proportion of patients do not attain remission. Major depressive disorder (MDD) bears several key neurobiological similarities with Alzheimer's Disease, namely cognitive deficits, impaired neuroplasticity, neurodegeneration, and neuroinflammation. Inducing neuroplasticity and reducing neuroinflammation are thought to be key cellular targets in the treatment of MDD. However, 40 Hz light stimulation research in the context of MDD is limited.

In this double-blinded, randomized placebo-controlled trial the primary objective is to investigate the antidepressant effect of a non-invasive neurostimulation therapy using a 40 Hz masked flickering light. This study utilizes a novel way of masking light by alternating the spectral composition of white light, resulting in the flicker unnoticeable to human perception.

The primary outcome measure of this study is the estimated difference in the Hamilton Depression Rating sub-scale (HAM-D6) scores between groups at week 6. Furthermore, investigators want to assess whether 40 Hz masked flickering light therapy produces a similar early shift in neural and cognitive response to emotional information seen with antidepressant therapy and whether this predicts treatment efficacy. Suicidal ideation, sleep patterns, and quality of life will be also investigated in order to evaluate the 40 Hz masked flickering light stimulation effects on other symptoms of depression. Explorative analysis of the EEG data will be performed from baseline to week 6 for the further development and validation of EEG-based biomarkers.

A total of 60 participants will be enrolled for a six weeks treatment period followed by a two weeks follow-up period. Participants will be recruited from a psychotherapeutic outpatient unit. Medication should be unchanged for the last 4 weeks and during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 18 and 75 years of age.
2. Subjects with a diagnosis of major depressive episode and currently experiencing a depressive episode according to DSM-5
3. Subjects with an MDI score > 21 at screening
4. Subjects on stable medication and/or psychotherapy for at least 4 weeks before starting the trial.
5. Subjects, who are willing to comply with the scheduled plan and are able to use the device for 1 hour per day for 6 weeks.
6. Subjects who can understand the oral and written study information and willing to sign an informed consent.

Exclusion Criteria:

1. Subjects with a history of photosensitive migraines and/or epileptic seizures
2. Subjects with a known eye disorder that might be sensitive to light treatment.
3. Subjects with a known history of bipolar disorder according to DSM-5 criteria
4. Subjects with suicidal ideation corresponding to a score of 2 or more on the HAM-D 17 scale item 3 or if the patient or investigator is uncertain of the degree of suicidal risk
5. Subjects with current psychotic symptoms. However, subjects with a prior psychotic depression or subjects with an actual psychotic depression episode that at the time of informed consent no longer fulfills the psychosis criteria are allowed to participate.
6. Subjects with current drug or alcohol dependence based on their medical records or the M.I.N.I. interview.
7. Subjects with a known history of borderline personality disorder
8. Subjects currently enrolled in another investigational treatment study.
9. Subjects with progressive neurodegenerative or neoplastic disease.
10. Subjects who are unable to understand the study procedures or handling of the NSS device.
11. Subjects who are pregnant at the time of inclusion or unsafe contraception in women of fertile age

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Depression severity measured by Hamilton Depression Rating sub-scale (HAM-D6) | Baseline and week 6
  The HAM-D6 scale is designed to rate the severity of depression by a healthcare professional. The assessment scale contains 6 items pertaining to the symptoms of depression experienced over the week. The primary endpoint is the mean difference in scores between treatments at baseline and week 6. The score range is from, 0-24 (24=highest depression level).

SECONDARY OUTCOMES:
Self-reported depression symptoms measured by Major Depression Inventory (MDI) | Baseline, week 1, 3, 6 and 8.
  The MDI is a depression self-assessment questionnaire. It consists of the 10 ICD-10 symptoms for depression. The sum of 10 questions indicates the degree of depression. The score range is from 0-50 (50=highest depression level).
Cognition measured by Facial Expression Recognition Test (FERT) | Baseline, week 1 and 6
  Assessing attention and recognition of emotional facial expressions using the FERT.
  The outcome is accuracy (% correct expressions identified, range: 0-100, higher is better) and response times for accurate identifications (milliseconds, range can vary quite a bit, smaller number is better because it reflect higher speed).
Cognition measured by Emotional Categorization and Memory test (ECMT) | Baseline, week 1 and 6
  Assessing self-referent memory for emotional words using the ECMT. Outcome is response times for correct identifications during encoding phase (milliseconds, smaller better) and for recall phase: number of positive and negative words recalled (higher is better)
Cognition measured by Screen for Cognitive Impairment in Psychiatry (SCIP) | Baseline, week 1 and 6
  Non-emotional cognition is investigated with the SCIP. Outcomes is total score as well as scores for the five subtests, in all cases higher is better (numbers correct)
Cognition measured by Trail Making Test B (TMT- B) | Baseline, week 1 and 6
  Non-emotional cognition investigated with the Trail Making Test B (TMT- B). Outcome is time in seconds to complete the task, lower is better (higher speed)
Sleep quality measured by Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 3, 6 and 8
  PSQI consist of seven component scores that are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A cut-off of 5 is recognized a indicative of sleep problems.
Sleep duration | Baseline, week 3, 6 and 8
  Average sleep duration assessed over last 7 days will be logged by the participants using a sleep diary.
Sleep timing | Baseline, week 3, 6 and 8
  Average sleep timing will be assessed over last 7 days logged by the participants using a sleep diary.
Quality of Life measured by WHO quality of life index (WHO-5) | Baseline, week 3,6 and 8
  The WHO-5 score ranges from 0 to 25, with 0 representing worst possible and 25 representing best possible quality of life. To obtain a percentage score ranging from 0 to 100, the raw score is multiplied by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life. A 10% difference indicates a significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Martiny, Principal Investigator — Senior Consultant at Psychiatric Centre Copenhagen
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agger MP, Carstensen MS, Henney MA, Hansen LS, Baandrup AO, Nguyen M, Petersen PM, Madsen KH, Kjaer TW. Novel Invisible Spectral Flicker Induces 40 Hz Neural Entrainment with Similar Spatial Distribution as 40 Hz Stroboscopic Light. J Alzheimers Dis. 2022;88(1):335-344. doi: 10.3233/JAD-220081. PMID 35570490
- [Background] Adaikkan C, Middleton SJ, Marco A, Pao PC, Mathys H, Kim DN, Gao F, Young JZ, Suk HJ, Boyden ES, McHugh TJ, Tsai LH. Gamma Entrainment Binds Higher-Order Brain Regions and Offers Neuroprotection. Neuron. 2019 Jun 5;102(5):929-943.e8. doi: 10.1016/j.neuron.2019.04.011. Epub 2019 May 7. PMID 31076275
- [Background] Chen X, Shi X, Wu Y, Zhou Z, Chen S, Han Y, Shan C. Gamma oscillations and application of 40-Hz audiovisual stimulation to improve brain function. Brain Behav. 2022 Dec;12(12):e2811. doi: 10.1002/brb3.2811. Epub 2022 Nov 14. PMID 36374520
- [Background] Cimenser A, Hempel E, Travers T, Strozewski N, Martin K, Malchano Z, Hajos M. Sensory-Evoked 40-Hz Gamma Oscillation Improves Sleep and Daily Living Activities in Alzheimer's Disease Patients. Front Syst Neurosci. 2021 Sep 24;15:746859. doi: 10.3389/fnsys.2021.746859. eCollection 2021. PMID 34630050
- [Background] Colgin LL, Moser EI. Gamma oscillations in the hippocampus. Physiology (Bethesda). 2010 Oct;25(5):319-29. doi: 10.1152/physiol.00021.2010. PMID 20940437
- [Background] Duman RS, Aghajanian GK, Sanacora G, Krystal JH. Synaptic plasticity and depression: new insights from stress and rapid-acting antidepressants. Nat Med. 2016 Mar;22(3):238-49. doi: 10.1038/nm.4050. PMID 26937618
- [Background] Fitzgerald PJ, Watson BO. Gamma oscillations as a biomarker for major depression: an emerging topic. Transl Psychiatry. 2018 Sep 4;8(1):177. doi: 10.1038/s41398-018-0239-y. PMID 30181587
- [Background] Godlewska BR, Harmer CJ. Cognitive neuropsychological theory of antidepressant action: a modern-day approach to depression and its treatment. Psychopharmacology (Berl). 2021 May;238(5):1265-1278. doi: 10.1007/s00213-019-05448-0. Epub 2020 Jan 15. PMID 31938879
- [Background] Martiny K, Lunde M, Unden M, Dam H, Bech P. Adjunctive bright light in non-seasonal major depression: results from clinician-rated depression scales. Acta Psychiatr Scand. 2005 Aug;112(2):117-25. doi: 10.1111/j.1600-0447.2005.00574.x. PMID 15992393